CLINICAL TRIAL: NCT03121885
Title: MetaboDyn- Liquid-liquid Extraction of Single Drops of Whole Capillary Blood as a Reliable Method of Measuring Metabolic Effects of Exercise: A Pilot Study.
Brief Title: Human Metabolic Dynamics at Rest and During Aerobic Exercise Under Normobaric Normoxic and Moderate Hypoxic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Gollasch (Other)
Collaborators: Max Delbrück Center for Molecular Medicine in the Helmholtz Association (MDC) Berlin (Unknown)
Responsible Party: Sponsor-Investigator, Benjamin Gollasch, Dr. med. Benjamin Gollasch, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MetaboDyn
Record Dates: First submitted 2017-03-31; First posted 2017-04-20 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2017-07

CONDITIONS: Energy Metabolism; Hypoxia; Metabolism and Nutrition Disorder
MeSH Terms: conditions — Hypoxia; Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: 30-minute movement activity — The subjects arrive in the CRU after a 12 hours overnight fast to perform a 30-minute movement activity with individually adapted exercise intensity on the treadmill.
Other: Hypoxia — The 30-minute movement activity on the treadmill will be completed by each subject once under normobaric normoxic and once under normobaric hypoxic conditions (equivalent to approximately 3000 meters above sea level) in a randomized episode.

SUMMARY:
The aim is to define in detail metabolic pathways at rest and during aerobic exercise in normal and healthy men and women under normobaric normoxic and moderate hypoxic conditions, using metabolomics technologies based on minimally invasive sampling relying on gas chromatography and mass spectrometry.

ELIGIBILITY:
Inclusion criteria:

* approval and written, informed consent
* healthy adults of varying fitness levels (age >18 years to 75 years)

Exclusion criteria:

* chronic illness requiring any medication
* pregnancy
* limitations regarding functioning in the hypoxic chamber
* inability to follow simple instructions
* relevant or severe abnormalities in medical history, physical examination, ECG routine laboratory parameters from blood and urine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of relative quantities of metabolites and physiological parameters related to its dynamic during exercise under normoxic and hypoxic conditions, using GC-MS. | 6 months
  A drop of capillary blood (20 µl) will be collected from the hyperemic earlobe for metabolomic analysis at the times t = 0 min (before starting), 10 min, 20 min and 30 min during the activity, and t = 50 and 60 min taken in the recovery phase. The oxygen saturation and heart rate will be determined at the same time points by pulse oximetry and heart rate monitoring, as well as blood gas analyses and subjective self-perception of energy availability on a quantitative scale throughout exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Experimental & Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Liquid-liquid extraction of single drops of whole capillary blood with collaborator partner MDC